CLINICAL TRIAL: NCT02236195
Title: An Open-Label, Single-Arm, Phase 2 Study of Mocetinostat in Selected Patients With Inactivating Alterations of Acetyltransferase Genes in Previously Treated Locally Advanced or Metastatic Urothelial Carcinoma
Brief Title: Study of Mocetinostat in Patients With Urothelial Carcinoma Having Inactivating Alterations of Specific Genes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-018
Record Dates: First submitted 2014-09-04; First posted 2014-09-10 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial; Bladder; HDAC; MGCD0103; Mocetinostat; CREBBP; EP300; Mirati; MethylGene
MeSH Terms: conditions — Carcinoma, Transitional Cell; Rubinstein-Taybi Syndrome | interventions — mocetinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mocetinostat (Experimental): Mocetinostat (MGCD0103) oral capsules three times weekly, 70 mg doses in first month, with increase to 90 mg doses if tolerated
  Interventions: Drug: Mocetinostat

INTERVENTIONS:
Drug: Mocetinostat
  Other Names: MGCD0103

SUMMARY:
Mocetinostat is an orally administered histone deacetylase (HDAC) inhibitor. This study is a Phase 2 trial evaluating the efficacy of mocetinostat in patients that have advanced urothelial carcinoma that has specific changes in tumor genes. Patients must have previously received treatment with chemotherapy that included a "platinum-containing agent" such as cisplatin. The study will enroll in stages, with 15 patients in the first stage. More patients will be added to the study if enough patients having beneficial responses are observed. Mocetinostat will be administered using oral capsules three times each week (eg, Monday, Wednesday and Friday). The study is designed to evaluate whether the number of patients responding to treatment is substantially higher than would be expected with other available treatments.

DETAILED DESCRIPTION:
To be eligible for this study, patient tumor testing must demonstrate a genetic alteration resulting in the loss of function of the Histone Acetyltransferase (HAT) family genes, CREBBP and/or EP300, including gene deletions or selected inactivating mutations. If testing has not already been performed, the study will provide for the testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of urothelial carcinoma
* Metastatic or locally advanced disease
* Prior chemotherapy that included a platinum agent
* Test results showing genetic change in tumor gene for CREBBP and/or EP300
* At least one tumor that can be measured

Exclusion Criteria:

* Uncontrolled tumor in the brain
* Impaired heart function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing tumor size reduction | Up to 4 months
  Tumors will be measured using radiographic scans. Tumor size reduction and overall disease response will be categorized according to the Response Evaluation Criteria In Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
Number of patients experiencing adverse events | Up to 12 months
Peak blood plasma concentration of mocetinostat | Up to 48 hours

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of Alabama, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Grivas P, Mortazavi A, Picus J, Hahn NM, Milowsky MI, Hart LL, Alva A, Bellmunt J, Pal SK, Bambury RM, O'Donnell PH, Gupta S, Guancial EA, Sonpavde GP, Faltaos D, Potvin D, Christensen JG, Chao RC, Rosenberg JE. Mocetinostat for patients with previously treated, locally advanced/metastatic urothelial carcinoma and inactivating alterations of acetyltransferase genes. Cancer. 2019 Feb 15;125(4):533-540. doi: 10.1002/cncr.31817. Epub 2018 Dec 20. PMID 30570744